CLINICAL TRIAL: NCT03768050
Title: Protocol for the Evaluation of Community-based Care for the Frail Elderly in Badalona Serveis Assistencials
Brief Title: Evaluation of Community-based Care for the Frail Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Roca, Consultor Senior, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SELFIE-BSA
Record Dates: First submitted 2018-11-28; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Chronic Disease; Frail Elderly Syndrome
Keywords: integrated care
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced care for frail elderly (Active Comparator): Integrated care program for frail elderly covering Home Hospitalization/Early Discharge; geriatric residences and; home-based case management done by dedicated teams specialised in geriatric medicine
  Interventions: Other: Advanced care for frail elderly
- Standard care (No Intervention): Usual care at the community and geriatric residences by primary care physicians

INTERVENTIONS:
Other: Advanced care for frail elderly — Home-based case management group receives advanced nursing care meeting the health and social needs of patient and/or carer. It is carried out through a process of evaluation, planning&coordination, facilitating the provision, monitoring and evaluation of the options and resources necessary for the resolution of the case. It is person-centred. The service also provides palliative care.
  Home hospitalisation/early discharge dispenses medical and nursing care at home on a transient basis after hospitalisation when patients still need surveillance and assistance. It is done in the acute, subacute or post-acute phase. In the last phase the focus is on functional recovery.
  The geriatric residences group is assisted by health care teams with expertise in geriatrics. They coordinate with primary care and health professionals of the residences to improve the attention. They are highly accessible, have high-resolutive capacity and can activate the resources of the healthcare network.
  Arms: Advanced care for frail elderly

SUMMARY:
The term frail chronic complex patient (CCP) is generally applied to subjects with heterogeneous conditions that may represent at least one of the following three traits: (i) the need for management by a number of specialists from different disciplines that often leads to high use of healthcare resources; (ii) fragility, which requires additional support either due to functional decline, social deficits and/or transient situations such as hospital discharge or, (iii) the need for highly specialised care with home technological support.

The current protocol deals with the second category of patients, frail CCP, and addresses horizontal integration of community-based services. It is based in the city of Badalona (216K inhabitants), within the metropolitan area of Barcelona. Badalona Serveis Assistencials (BSA) is the service provider of integrated care services for this population.

DETAILED DESCRIPTION:
The study will assess three types of specific groups of patients: (i) Early discharge group includes patients acutely admitted to the medical and/or surgical hospital wards and promptly discharged to receive home-based post-acute care and/or rehabilitation; (ii) Home-based Case Management group includes complex chronic patients or patients receiving long-term care by a case management nurse; and (iii) Geriatric residences group will include patients receiving acute support, post-acute or continued care for elderly people living in geriatric residences.

It will be conducted by Badalona Serveis Assistencials (BSA), an integrated care service provider located in the city of Badalona (420K inhabitants) in the North-Eastern part of the Barcelona Metropolitan Area.

The current study protocol aims to assess cost-effectiveness of the three types of interventions for frail patients, as well as to generate a roadmap for regional scalability of the service. The study design will consist of a prospective quasi-experimental case-control design wherein each intervention group will be compared with the corresponding usual care group (controls, 1:1 ratio), using propensity score matching. Age, sex, GMA (adjusted morbidity groups), socioeconomic status, number of hospitalisations during the previous year and polypharmacy will be used as matching variables.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 65 years.
* Complexity: ≥ 2 chronic diseases
* Polypharmacy: ≥ 4 drugs
* Registered as complex chronic patient
* ≥ 3 hospital or emergency room readmissions in the last year
* Having suffered a recent acute illness requiring continuous clinical and/or rehabilitative care by the Home Hospitalisation Unit or primary care.
* To be admitted in one of the geriatric residences of the territory of Badalona, Montgat and Tiana.

Exclusion criteria

* Any neurological disease (e.g. severe-phase dementia with global deterioration scale (GDS) ≥ 7) or psychiatrically severe enough not to allow the subject to respond to questionnaires.
* Subjects who do not agree to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Costs | 30 days
  Health Care Costs

SECONDARY OUTCOMES:
Number of hospital admissions | 30 days
  Number of hospital admissions during the study period
Patient centred healthcare provision | 30 days
  Patient centred healthcare provision as measured by the Person Centred Coordinated Experience Questionnaire
Continuity of care within the healthcare system | 30 days
  Continuity of care within the healthcare system as measured by the Nijmegen Continuity of Care Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Josep Roca, MD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NEXTCARE is an innovation project belonging to the Healthcare Ris3Cat community lead by Biocat which officially starts on October 2016 — http://www.nextcarecat.cat
- See also: SELFIE (Sustainable intEgrated care modeLs for multi-morbidity: delivery, FInancing and performancE) is a Horizon2020 European Union project — http://www.selfie2020.eu/